CLINICAL TRIAL: NCT04658524
Title: Evaluation of Thyroid Function in Patients With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rio de Janeiro State University (Other)
Responsible Party: Principal Investigator, Ana Beatriz Winter Tavares, Professor, Rio de Janeiro State University
Other Study IDs: 3.138.270
Record Dates: First submitted 2020-11-20; First posted 2020-12-08 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Chronic Kidney Disease; Thyroid Dysfunction
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Thyroid Function Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chonic kidney disease stages 3, 4 and 5: Patients with stage chronic kidney disease stages 3, 4 and 5. CKD stages were defined according to the Kidney Disease Improving Global Outcomes directives (KDIGO): a) stage 3A: eGFR 45 and 59 ml/min/1.73m2; b) stage 3B: eGFR between 30 and 44 ml/min/1.73m2; c) stage 4: eGFR between 15 and 29 ml/min/1.73 m2
  Interventions: Diagnostic Test: Thyroid function

INTERVENTIONS:
Diagnostic Test: Thyroid function — laboratorial thyroid tests

SUMMARY:
A higher prevalence of thyroid disease has been associated with chronic kidney disease (CKD), and subclinical hypothyroidism seems to be the most common dysfunction. The aim is to evaluate thyroid function and autoimmunity in patients with CKD stages 3, 4 and 5. Cross-sectional study to be carried out on patients with stages 3 and 4 in a Nephrology outpatient clinic. Thyroid function is evaluated by measuring thyroid stimulating hormone (TSH), free thyroxine, free triiodothyronine and antithyroperoxidase antibodies (TPOAb) levels.

DETAILED DESCRIPTION:
Cross-sectional study to be carried out on patients with stages 3, 4 and 5 in a Nephrology outpatient clinic. Thyroid function is evaluated by measuring thyroid stimulating hormone (TSH), free thyroxine, free triiodothyronine and antithyroperoxidase antibodies (TPOAb) levels. Free Thyroxine (FT4) will be measured by liquid chromatography tandem mass spectrometry and electrochemiluminescence immunoassay in order to compare methods in this population.

The glomerular filtration rate was estimated (eGFR) by the Chronic Kidney Disease Epidemiology Collaboration formula (CKD-EPI), and the CKD stages were defined according to the Kidney Disease Improving Global Outcomes directives (KDIGO).

ELIGIBILITY:
Inclusion Criteria:Patients over 18 years old with CKD stages 3 and 4 were included in the study.

-

Exclusion Criteria: 1) acute systemic inflammatory disease; 2) pituitary disease in the past or present; 3) regular treatment with amiodarone, lithium, interferon, immunosuppressive drugs and glucocorticoids; 4) previously diagnosed hypothyroidism and undergoing levothyroxine replacement.

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Chronic kidney disease patients followed in a Nephrology outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Free thyroxine (FT4) levels in chronic kidney disease | through study completion, an average of 3 years
  Free thyroxine levels through two different methods
TSH levels in chronic kidney disease | through study completion, an average of 3 years
  TSH levels

SECONDARY OUTCOMES:
Frequency of thyroid antibodies in chronic kidney disease | through study completion, an average of 3 years
  antithyroperoxidase and antitireoglobulin antibodies
Free triiodothyronine (FT3) levels in chronic kidney disease | through study completion, an average of 3 years
  T3 levels

CONTACTS AND LOCATIONS:
Locations (1):
- Ana Beatriz Winter Tavares, Petrópolis, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhee CM. The interaction between thyroid and kidney disease: an overview of the evidence. Curr Opin Endocrinol Diabetes Obes. 2016 Oct;23(5):407-15. doi: 10.1097/MED.0000000000000275. PMID 27428519
- [Background] Mariani LH, Berns JS. The renal manifestations of thyroid disease. J Am Soc Nephrol. 2012 Jan;23(1):22-6. doi: 10.1681/ASN.2010070766. Epub 2011 Oct 21. PMID 22021708
- [Background] Meuwese CL, Gussekloo J, de Craen AJ, Dekker FW, den Elzen WP. Thyroid status and renal function in older persons in the general population. J Clin Endocrinol Metab. 2014 Aug;99(8):2689-96. doi: 10.1210/jc.2013-3778. Epub 2014 Apr 15. PMID 24735423
- [Derived] Scandelai KS, Vianna PDBFA, Sanches JPB, Bregman R, Tavares ABW. Correlation between thyroid function and proteinuria in patients with chronic kidney disease stages 3 and 4. Int Urol Nephrol. 2025 Dec;57(12):4309-4314. doi: 10.1007/s11255-025-04646-4. Epub 2025 Jul 5. PMID 40615656